CLINICAL TRIAL: NCT01770899
Title: A Prospective Analysis of the Use of Oral Montelukast in Children With Status Asthmaticus
Brief Title: Evaluation Montelukast in the Treatment of Status Asthmaticus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Corrie Fletcher (Other)
Responsible Party: Sponsor-Investigator, Corrie Fletcher, Pediatric Resident, Advocate Center for Pediatric Research
Organization: Advocate Center for Pediatric Research (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5441
Record Dates: First submitted 2013-01-15; First posted 2013-01-18 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Status Asthmaticus
Keywords: Montelukast; Singulair; status asthmaticus
MeSH Terms: conditions — Status Asthmaticus | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Montelukast (Experimental): Montelukast 5mg capsules for 2-5 year old every 24h and 8mg capsules for 6-14 year olds every 24h.
  Interventions: Drug: Montelukast
- Placebo (Placebo Comparator): One placebo capsule given every 24h
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Montelukast
  Other Names: Singulair
  Arms: Montelukast
Drug: Placebo — Gelatin capsule given every 24 hours
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effectiveness of oral montelukast (Singulair) given with other standard asthma medications and treatments in the treatment of children with status asthmaticus. Status asthmaticus is an acute asthma attack that does not respond to standard intermittent treatments but requires a continuous medication to aid in breathing. While new medications have been used to better manage chronic asthma, acute asthma exacerbations continue to be a significant cause of hospitalization and even death in children. Oral montelukast is a very safe medication that is used to manage chronic asthma in children, but it has not been studied for use in status asthmaticus. If oral montelukast, given with other standard therapies, can reduce the treatment length associated with severe, acute asthma exacerbations in children, it could potentially improve both the morbidity and burden of pediatric asthma.

DETAILED DESCRIPTION:
While new medications have been used to better manage chronic asthma, acute exacerbations continue to be a significant cause of pediatric morbidity and mortality. Montelukast holds an established role in the pediatric outpatient management of asthma and while two promising studies in adults have demonstrated its potential use as an adjunctive therapy for acute exacerbations, its similar use in pediatrics has yet to be established. This pilot study is designed as a prospective, double blinded, randomized, controlled, clinical trial comparing the use of oral montelukast plus standard of care vs. standard of care alone in children admitted for status asthmaticus to the pediatric intensive care unit (PICU). The primary outcome the investigators are interested in is the time to reach a Modified Pediatric Asthma Score (PAS) of < 5, which, per the clinical protocol for the treatment of status asthmaticus, is the time when patients are able to come off continuous bronchodilator therapy. If oral montelukast, given with other standard therapies, can reduce the treatment, emotional, and financial burden (e.g., shortened intensive care stay) associated with severe, acute asthma exacerbations in children, it would provide a significant therapeutic advantage, potentially improving both the morbidity and burden of pediatric asthma.

ELIGIBILITY:
Inclusion criteria:

* Between ages 2-148 years
* Requiring PICU admission for status asthmaticus
* Able to take oral medication
* Pediatric asthma score > 8 on admission

Exclusion criteria:

* Intubated patients or other patients unable to take medications by mouth secondary to anatomic or pre-existing craniofacial issues
* Patients already on montelukast as their controller medication
* Patients with a known allergy to montelukast
* Any patient with phenylketonuria (PKU)
* Any patient currently on treatment with rifampin, fluconazole, or Phenobarbital medications

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2013-01; Primary Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Improvement of pediatric asthma score | Hourly during the length of the patient's pediatric ICU hospitalization for status asthmaticus
  Measurement of pediatric asthma score hourly from admission assessing for time to improvement of score, an average length of stay predicted 2-4 days.

CONTACTS AND LOCATIONS:
Overall Officials: Corrie Fletcher, DO, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Advocate Children's Hospital Oak Lawn, Oak Lawn, Illinois, United States